CLINICAL TRIAL: NCT02640573
Title: Treatment of Adult Patients With Hemoglobin SC Disease
Brief Title: Treatment of Adult Patients With Hemoglobin SC Disease (SCYTHE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Baylor College of Medicine (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Vivien Sheehan, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37290 IM-SCYTHE
Record Dates: First submitted 2015-12-17; First posted 2015-12-29 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hemoglobin SC Disease
MeSH Terms: conditions — Hemoglobin SC Disease | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (1):
- Hydroxurea (Experimental): Initiate hydroxyurea at 10 mg/kg daily and escalate hydroxyurea dose by 5 mg/kg/day every 8 weeks up to a maximum dose of 35 mg/kg/day if blood counts meet escalation criteria.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Treat symptomatic HbSC patients to MTD on hydroxyurea, and assess for clinical improvement using the AdultsQLTM 3.0 Sickle Cell Disease Module after 6 months at MTD, compared to entrance scores

SUMMARY:
Sickle cell disease (SCD), specifically hemoglobin SC disease (HbSC), is a subtype of sickle cell disease with typically higher hemoglobin and milder or later disease complications. Sickle cell disease is a disorder in which red blood cells (RBCs) are abnormally shaped. This can result in painful episodes, serious infections, and damage to body organs. One medication used to treat sickle cell disease is hydroxyurea.

Hydroxyurea therapy offers significant benefits for infants, children, and adolescents with sickle cell anemia. These include a reduction in the frequency of pain crises and acute chest syndrome (inflammation of the lungs). Hydroxyurea has been given to many HbSC patients but HbSC patients were not included in the large clinical trials used to test hydroxyurea in SCD, so less is known about how HbSC patients respond to hydroxyurea.

The purpose of this research study is to see if hydroxyurea, a medication given to many patients with the most common type of sickle cell, those who are homozygous for the sickle mutation (HbSS), helps individuals who have HbSC. The investigators will see if it helps by giving a questionaire when the medication is started, and then every two months at a clinic visit. The questionaire, called the AdultsQLTM 3.0 Sickle Cell Disease Module, measures quality of life. The investigators will also see how hydroxyurea changes laboratory test numbers, and blood thickness.

DETAILED DESCRIPTION:
Patients will be recruited from the patient population followed at the Texas Children's Cancer and Hematology Centers (TCC/HC)/Baylor College of Medicine (BCM) and the University of Texas Houston Hematology Center. To be eligible to participate in this study, patients must have HbSC disease, have experienced a sickle cell disease related complication, or have a score of 80 or lower on the AdultQLTM Sickle Cell Disease Module 3.0. This questionnaire will be offered to all patients with HbSC seen in our clinic that consent to this study. Patients must also agree to clinic visits every two months, and to phlebotomy, or blood removal after 6 months on the study if they meet criteria for phlebotomy.

If the patient is a sexually active female, they will be offered birth control. If the patient chooses not to initiate effective birth control, they will be tested at their scheduled visit with a urine pregnancy test. If the patient becomes pregnant they will be removed from the study.

Patients will be assessed in clinic every two months after starting treatment. Hydroxyurea will be started at 10 mg/kg/day, and increased by 5 mg/kg/day if needed to a maximum tolerated dose (MTD) of 35/mg/day. The most common side effect of the drug is a drop in infection fighting cells, or white blood cells, so the medication will be started at a low dose and the dose will be increased only if it is safe to do so. After 6 months at MTD on the study, patients will be evaluated for their response to hydroxyurea. If they have not reached their MTD after 6 months their time on the study will be increased to allow for 6 months observation at MTD. The minimum time the patients will be on the study is 12 months after starting hydroxyurea therapy with an option to participate in a 2 year observation study following the end of the study.

If the patients have had minimal or no benefit from the medication, monthly phlebotomy will be added to their treatment regimen, at 7-10 ml/kg. The first phlebotomy volume will be 7 ml/kg, but may be increased to 10 ml/kg to obtain the target Hb of 9-10 g/dL. Patients will remain on hydroxyurea and phlebotomy for six months. If their Hb is less than or equal to 9.0 g/dL on their phlebotomy visit, phlebotomy will not be performed and their phlebotomy visits will be spaced every 2 months. Patients time on the study will be increased to allow for 6 months observation to ensure that there is no late harmful effects. The minimum time patients will be on the study is 18 months after starting phlebotomy with an option to participate in a 2 year observation study following the end of the study.

Patients will be asked to allow the investigators to review information from their medical records at the start of the study, and throughout the study. If the patient would like to participate in the two year follow-up, their records will be reviewed during that period as well.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HbSC disease
* Score of 80 or lower on the AdultQLTM 3.0 Sickle Cell Disease Module, or any disease related complication, including, but not limited to, one or more pain events per year, proliferative sickle retinopathy, avascular necrosis, cholelithiasis, or any thrombotic event. If the subject has a score >80, they may still enroll on the trial, and be analyzed for secondary endpoints. They will be excluded from analysis of the primary endpoint.

Exclusion Criteria:

* Failure to meet inclusion criteria
* Hydroxyurea usage in the last 3 months.
* Chronic RBC transfusion therapy
* Packed red blood cell transfusion in the last 3 months (temporary exclusion).
* Pregnancy, or refusal to use medically effective birth control if female and sexually active.
* Current phlebotomy therapy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Sheehan, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxurea
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hydroxurea
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants] — chart review
  Participants
    <=18 years | 0
    Between 18 and 65 years | 1
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1
Fetal hemoglobin level at baseline [Mean (Full Range); unit: %] | 2 [2 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Fetal Hemoglobin Response to HU
Description: Change in HbF on hydroxyurea from baseline
Time Frame: Baseline to 6 months
Population: Baseline QoL only; no subsequent values obtained.
Groups:
- Single Arm Study: adult patient on HU, measure of QoL
Arm/Group | Single Arm Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Hydroxurea
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT02640573/Prot_SAP_000.pdf